CLINICAL TRIAL: NCT03187119
Title: Take Action for Asthma Control Study - Pilot Randomized Controlled Trial of Pictorial Asthma Action Plans to Promote Self-management and Health in Rural Youth With Asthma
Brief Title: Investigation of the Role of Pictorial Asthma Action Plans to Promote Self-management in Rural Youth With Asthma
Acronym: TAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Christina Duncan, Principal Investigator, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1612396282
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Pediatric; Education; Technology-supported intervention; Asthma Action Plan; Health literacy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pictorial Asthma Action Plan (Experimental): Young people in the Pictorial Asthma Action Plan (PAAP) arm will receive a PAAP generated by their asthma provider using a software program developed for the study. The PAAP will be personalized according to the young person's gender, race, favorite sport/activity, provider's gender, provider's clinic contact details, and hospital in emergency situations. The PAAP contains minimal text, instead illustrating each participant's asthma regimen using pictures, such as color-coded daily controller and rescue inhalers. Each participant will receive multiple copies of their PAAP, after receiving a brief education session with their provider, outlining the treatment summarized in the PAAP.
  Interventions: Behavioral: Pictorial Asthma Action Plan
- Written Asthma Action Plan (Active Comparator): Young people in the Written Asthma Action Plan (WAAP) arm will receive a WAAP generated by their asthma provider using using the National Heart, Lung, and Blood Institute (NHLBI) template. The WAAP will be personalized according to the young person's treatment plan. Each participant will receive multiple copies of their WAAP, after receiving a brief education session with their provider, outlining the treatment summarized in the WAAP.
  Interventions: Behavioral: Written Asthma Action Plan

INTERVENTIONS:
Behavioral: Pictorial Asthma Action Plan — Participants will receive a PAAP plan, personalized to their asthma treatment. Each participant will take part in a brief education session during which their asthma provider will outline the treatment plan summarized in their PAAP.
  Arms: Pictorial Asthma Action Plan
Behavioral: Written Asthma Action Plan — Participants will receive a WAAP plan, personalized to their asthma treatment. Each participant will take part in a brief education session during which their asthma provider will outline the treatment plan summarized in their WAAP.
  Arms: Written Asthma Action Plan

SUMMARY:
The aim of this study is to investigate the potential benefit of Pictorial versus Written Asthma Action Plans (AAPs) to support asthma management among young people with persistent asthma. Participants will be randomly allocated to the Pictorial or Written AAP group and followed up over a 6-month period. Qualitative and quantitative data will be collected from young people, parents and clinical teams involved in recruitment to assess the feasibility and acceptability of the Pictorial AAP (PAAP) software developed for this study, the PAAPs produced by the software, and the study procedures.

DETAILED DESCRIPTION:
Asthma is the most common chronic health condition of childhood, and continues to be associated with morbidity and mortality. Many children with persistent asthma follow a treatment plan including a prescription to take a daily inhaled corticosteroid (controller), often in conjunction with a daily oral controller medication, and a dose of an albuterol (rescue) inhaler before activity or exercise. Young people with asthma must add to this treatment plan in response to a flare in symptoms by taking additional medication and contacting their asthma provider or getting to a hospital. Adherence to daily medications is essential for maintaining lung health and reducing symptom flares, but asthma treatment is complex, requiring regular decision-making in response to symptoms and environmental issues like symptom triggers. As a result consistent adherence is a challenge for families and young people. It is recommended to provide an Asthma Action Plan (AAP) to all people diagnosed with asthma, summarizing their treatment plan using a traffic light format; Green Zone for daily, symptom-free management, Yellow Zone for symptom flare, and Red Zone for extreme symptom flare. Despite evidence for the effectiveness of AAPs, they are often not prescribed for reasons including readability and accessibility for families and young people, and asthma provider perceptions of their utility and suitability. In this study, young people with persistent asthma will be given a Written (WAAP) or Pictorial Asthma Action Plan (PAAP) to compare the differential impact on AAP knowledge, adherence to daily inhaler use, and asthma control. Software developed for the study, in collaboration with providers, young people with asthma and their parents, will be used to generate personalized PAAPs. Quantitative and qualitative data will be collected to explore perceptions of providers, parents and young people of different versions of AAPs, the influence of AAPs on asthma understanding and management, and the experience of taking part in the study, as well as to assess the impact of different AAPs on the asthma and psychosocial outcomes mentioned. The findings will inform the development of the PAAP software and as the basis for a definitive Randomized Controlled Trial of the efficacy of PAAPs.

ELIGIBILITY:
Inclusion Criteria:

* age 8-17 years
* new patient (to clinic) with a diagnosis of persistent asthma or an established patient with uncontrolled persistent asthma and a clinical need for a new treatment regimen
* no history of having received a written AAP
* prescribed an inhaled corticosteroid (i.e., daily controller medication).

Exclusion Criteria:

* patients and caregivers who do not use English as their primary language
* has a significant developmental (e.g., autism, intellectual disability) or sensory (e.g., blindness) disorder that would preclude completion of study measures.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Duncan, PhD, Principal Investigator — West Virginia University
Locations (1):
- WVU Medicine, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Started | 22 | 23
Completed | 20 | 18
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: The analysis population is the same from the assignment in Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 23 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.70 (2.91) | 11.87 (2.65) | 11.79 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 22 | 43
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45
Caregiver Age [Mean (Standard Deviation); unit: years] | 40.00 (7.92) | 42.26 (9.88) | 41.16 (8.95)
Parental Education [Count of Participants; unit: Participants]
  Mother: Less than High School | 3 | 7 | 10
  Mother: More than High School | 19 | 16 | 35
  Father: Less than High School | 7 | 11 | 18
  Father: More than High School | 15 | 12 | 27
Caregiver Marital Status [Count of Participants; unit: Participants] — Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., incomplete measures).
  Participants
    number analyzed (Participants) | 21 | 21 | 42
    Never Been Married / Single | 2 | 0 | 2
    Married to other biological parent | 14 | 13 | 27
    Living with boyfriend / girlfriend | 1 | 2 | 3
    Divorced / Single | 0 | 4 | 4
    Remarried to step-parent | 3 | 2 | 5
    Widowed (other biological parent is deceased) | 1 | 0 | 1
Annual Household Income [Count of Participants; unit: Participants] — Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., incomplete measures).
  Participants
    number analyzed (Participants) | 22 | 22 | 44
    Less than $15,000 | 3 | 2 | 5
    15,000 - $29,999 | 2 | 6 | 8
    $30,000 - $44,999 | 5 | 3 | 8
    $45,000 - $59,999 | 2 | 1 | 3
    $60,000 - $74,999 | 1 | 4 | 5
    $75,000 and greater | 9 | 6 | 15
Child Prior Diagnosis of Asthma [Count of Participants; unit: Participants]
  Yes | 20 | 19 | 39
  No | 2 | 4 | 6
Child Age of Diagnosis of Asthma [Mean (Standard Deviation); unit: years] — Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., equipment).
  years
    number analyzed (Participants) | 18 | 19 | 37
    (all) | 3.94 (2.93) | 7.30 (1.38) | 5.67 (4.07)
Child Number of Relatives with Asthma Diagnosis [Count of Participants; unit: Participants]
  Yes | 18 | 19 | 37
  No | 4 | 4 | 8
Child Immediate Relatives Asthma [Count of Participants; unit: Participants]
  Yes | 13 | 15 | 28
  No | 9 | 8 | 17
Child Extended Relatives Asthma [Count of Participants; unit: Participants]
  Yes | 13 | 16 | 29
  No | 9 | 7 | 16
Child Grade [Count of Participants; unit: Participants]
  Elementary (1-4) | 7 | 6 | 13
  Middle (5-8) | 9 | 12 | 21
  High (9-12) | 6 | 5 | 11
Child Special Education [Count of Participants; unit: Participants]
  Yes | 4 | 7 | 11
  No | 18 | 16 | 34
Child Illness Comorbidity [Count of Participants; unit: Participants]
  Yes | 16 | 11 | 27
  No | 6 | 12 | 18
Child Insurance Provider [Count of Participants; unit: Participants] — Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., incomplete measures).
  Participants
    number analyzed (Participants) | 21 | 21 | 42
    Medicaid | 19 | 18 | 37
    Private | 2 | 3 | 5
    None | 0 | 0 | 0
Asthma Control Test [Count of Participants; unit: Participants] — Asthma control was measures via the Asthma Control Test (ACT) 12 for participants 12 and older (Nathan et al., 2004), and the ACT 11 for participants 11 and younger (Liu et al., 2007). These scales include Likert type response options that differ by item, but for all items higher scores indicate more control. The raw scores were dichotomized for a clinical cut-off, with a score of 19 and less considered "poor control".
  Participants
    Above Clinical Cut Off (>19) | 11 | 7 | 18
    Below Clinical Cut Off (>19) | 11 | 16 | 27
Forced Expiratory Volume (FEV)1 [Mean (Standard Deviation); unit: percentage of predicted FEV1 value] — Lung function was assessed using spirometry outcome of Forced Expiratory Volume (FEV1). Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., equipment).
  percentage of predicted FEV1 value
    number analyzed (Participants) | 18 | 15 | 33
    (all) | 2.39 (0.86) | 2.32 (0.62) | 2.36 (0.75)
Forced Expiratory Flow (FEF) 25-75 [Mean (Standard Deviation); unit: percent predicted] — This data is gathered from a spirometry test. FEF 25-75 is the air flow between 25% and 75% of forced vital capacity.
  percent predicted | 2.29 (0.95) | 2.26 (0.68) | 2.28 (0.81)
The Asthma Action Plan Knowledge Interview (AAPKI)-Parent [Mean (Standard Deviation); unit: Average percent correct] — The Asthma Action Plan Knowledge Interview (AAPKI) was developed for the purposes of this study. The first section of the structured interview included 8 items that were scored as correct (1) or incorrect (0). Two items were excluded because they were not relevant to all participants. The second section of the structured interview included 3 open response on a 4-point scale: 0 = incorrect; 1 = possibly correct, but vague or missing important details; 2 = correct but not detailed; 3 = correct and specific. Percent correct knowledge scores were calculated for the nine questions.
  Average percent correct | 72.72 (17.39) | 71.50 (14.14) | 72.10 (15.65)
The Asthma Action Plan Knowledge Interview (AAPKI)-Child [Mean (Standard Deviation); unit: Average percent correct] — The Asthma Action Plan Knowledge Interview (AAPKI) was developed for the purposes of this study. The first section of the structured interview included 8 items that were scored as correct (1) or incorrect (0). Two items were excluded because they were not relevant to all participants. The second section of the structured interview included 3 open response on a 4-point scale: 0 = incorrect; 1 = possibly correct, but vague or missing important details; 2 = correct but not detailed; 3 = correct and specific. Percent correct knowledge scores were calculated for the nine questions.
  Average percent correct | 73.73 (17.67) | 58.94 (19.66) | 66.17 (19.95)
Wechsler Individual Achievement Test-III [Mean (Standard Deviation); unit: age-based percentile rank] — Wechsler Individual Achievement Test-III (WIAT-III) - Reading Comprehension subtest. This subtest is a measure of reading comprehension that is widely validated for use in children and adolescents. Participants' raw score on the WIAT-III will be converted age-based percentile rank.
  age-based percentile rank | 97.14 (10.8) | 95.22 (22) | 96.16 (17.25)
Test of Functional Health Literacy in Adults (TOFHLA) [Median (Inter-Quartile Range); unit: units on a scale] — The Short Test of Functional Health Literacy in Adults (S-TOFHLA) is a measure of a respondent's ability to read and understand health-related information. Each item is scored 1 for correct and 0 for incorrect. There is a total of 36 items. Scores range from 0-36. Total raw scores < 16 are reflective of "inadequate" literacy.
  units on a scale | 35 [35 to 35] | 35 [35 to 36] | 35 [35 to 35]
Test of Functional Health Literacy (Child) [Median (Inter-Quartile Range); unit: units on a scale] — The Short Test of Functional Health Literacy in Adults (S-TOFHLA) is a measure of a respondent's ability to read and understand health-related information. Each item is scored 1 for correct and 0 for incorrect. There is a total of 36 items. Scores range from 0-36. Total raw scores < 16 are reflective of "inadequate" literacy. The measure was only administered to participants aged 13-17, as the measure has been validated in this age group, but not with younger children. Population: The number of cases analyzed differed from the overall number analyzed due to some participants below age cutoff.
  units on a scale
    number analyzed (Participants) | 8 | 10 | 18
    (all) | 34.5 [33 to 35] | 34 [32 to 35] | 34 [32 to 35]
Asthma Numeracy Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — The Asthma Numeracy Questionnaire (ANQ) assessed specific numerical skills used in asthma self-management. It is a 4-item questionnaire of numerical concepts (arithmetic and percentage) adapted from standard asthma education (Apter et al., 2006).The score is the number correct and ranges from 0 to 4. Lower scores indicate lower asthma numeracy. Higher scores indicates higher asthma numeracy.
  units on a scale | 3.5 [3 to 4] | 4 [3 to 4] | 4 [3 to 4]

OUTCOME MEASURES:

1. Primary Outcome: The Asthma Action Plan Knowledge Interview (AAPKI)-Child
Description: The Asthma Action Plan Knowledge Interview (AAPKI) was developed for the purposes of this study. The first section of the structured interview included 8 items describing hypothetical situations in which the respondent was asked to categorize themselves or their child into one of three zones. These items were scored as correct (1) or incorrect (0). Two items were excluded because they were not relevant to all participants. The second section of the structured interview included 3 open response items asking the respondent to describe the treatment instructions for the three zones according to the AAP. Responses were coded on a 4-point scale: 0 = incorrect; 1 = possibly correct, but vague or missing important details; 2 = correct but not detailed; 3 = correct and specific. Percent correct knowledge scores were calculated using six items from the first section and the three additional questions about treatment, for a total of nine questions.
Time Frame: Measured at three time points over 6 months; baseline, 3- and 6-month follow-up.
Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., attrition, incomplete measures).
Measure: Mean (Standard Error); unit: Average Percent Correct
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 23
Average Percent Correct
  3 Month Assessment: number analyzed (Participants) | 19 | 18
  3 Month Assessment | 76.11 (20.16) | 61.40 (11.33)
  6 Month Assessment: number analyzed (Participants) | 15 | 17
  6 Month Assessment | 77.08 (17.90) | 62.09 (11.15)
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this model is the Pictorial Asthma Action Plan Group; Test type: Superiority; p = 0.42, linear mixed model — The results listed here are for the main effect of time. Please see Analyses 2 and 3 for the main effect of group and the time x group interaction; Slope = 1.41
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.03, multiple linear regression. — The results listed here are for the main effect of group. Please see Analyses 1 and 3 for the main effect of time and the time x group interaction; Slope = -14.31
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.89, multiple linear regression. — The results listed here are for the time x group interaction. Please see Analyses 1 and 2 for the main effects of group and time; Slope = -0.33

2. Primary Outcome: The Asthma Action Plan Knowledge Interview (AAPKI)-Parent
Description: The Asthma Action Plan Knowledge Interview (AAPKI) was developed for the purposes of this study. The first section of the structured interview included 8 items describing hypothetical situations in which the respondent was asked to categorize their child into one of three zones. These items were scored as correct (1) or incorrect (0). Two items were excluded because they were not relevant to all participants. The second section of the structured interview included 3 open response items asking the respondent to describe the treatment instructions for the three zones according to the AAP. Responses were coded on a 4-point scale: 0 = incorrect; 1 = possibly correct, but vague or missing important details; 2 = correct but not detailed; 3 = correct and specific. Percent correct knowledge scores were calculated using six items from the first section and the three additional questions about treatment, for a total of nine questions.
Time Frame: Measured at three time points over 6 months; baseline, 3- and 6-month follow-up.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average Percent Correct
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 23
Average Percent Correct
  3 Month Assessment: number analyzed (Participants) | 19 | 18
  3 Month Assessment | 74.44 (16.95) | 69.59 (13.78)
  6 Month Assessment: number analyzed (Participants) | 15 | 14
  6 Month Assessment | 63.89 (14.91) | 65.28 (10.64)
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.31, multiple linear regression. — [p-value comment as in outcome 1, analysis 1]; Slope = -1.59
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.73, multiple linear regression. — [p-value comment as in outcome 1, analysis 2]; Slope = 1.90
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.92, multiple linear regression. — [p-value comment as in outcome 1, analysis 3]; Slope = -0.21

3. Primary Outcome: Asthma Control Test
Description: Asthma control was measures via the Asthma Control Test (ACT) 12 for participants 12 and older (7 items), and the ACT 11 for participants 11 and younger (5 items). These scales include a 5 point Likert type response. Total score is calculated by summing response with higher scores indicating more control. Possible range of scores is 0-35. The raw scores were dichotomized for a clinical cut-off, with a score of 19 and less considered "poor control".
Time Frame: Measured at four time points over 6 months; baseline, 1-, 3- and 6-month follow-up.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 23
Participants
  1 Month Assessment: number analyzed (Participants) | 22 | 22
  1 Month Assessment: Above ACT cut-off (>19) | 19 | 11
  1 Month Assessment: Below ACT cut-off (>19) | 3 | 11
  3 Month Assessment: number analyzed (Participants) | 20 | 19
  3 Month Assessment: Above ACT cut-off (>19) | 17 | 16
  3 Month Assessment: Below ACT cut-off (>19) | 3 | 3
  6 Month Assessment: number analyzed (Participants) | 16 | 17
  6 Month Assessment: Above ACT cut-off (>19) | 12 | 13
  6 Month Assessment: Below ACT cut-off (>19) | 4 | 4
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.06, generalized linear mixed model — [p-value comment as in outcome 1, analysis 1]; Slope = 0.52
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.07, generalized linear mixed model — The results listed here are for the main effect of group. Please see Analyses 1 and 2 for the main effect of group and the time x group interaction; Slope = -1.57
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.33, generalized linear mixed model — The results listed here are for the time x group interaction. Please see Analyses 2 and 3 for the main effects of group and time; Slope = 0.37

4. Primary Outcome: Adherence to Daily Controller Inhaler
Description: Adherence to daily controller inhaler measured objectively using an electronic monitor attached to the inhaler and connected to a smart phone application or 'hub' in the participant's home.Data was examined for daily percent adherence by comparing the number of puffs taken with the number of puffs prescribed. Day 180 was not included in the analyses due to low insufficient group size.
Time Frame: Measured over 6 months; day 1, day 30, day 90 and day 180
Population: For this pilot program, prescription dose was not used for randomization into group. Only one participant had 1 puff per day; all other participants had 2 or 4. Thus, this participant taking only one per day was excluded from adherence analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of daily adherence
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 21 | 23
percentage of daily adherence
  Day 1: 2x per day prescription: number analyzed (Participants) | 10 | 6
  Day 1: 2x per day prescription | 50 [50 to 100] | 75 [50 to 100]
  Day 1: 4x per day prescription: number analyzed (Participants) | 11 | 17
  Day 1: 4x per day prescription | 50 [50 to 75] | 50 [50 to 75]
  Day 30: 2x per day prescription: number analyzed (Participants) | 10 | 5
  Day 30: 2x per day prescription | 50 [50 to 100] | 100 [100 to 100]
  Day 30: 4x per day prescription: number analyzed (Participants) | 10 | 16
  Day 30: 4x per day prescription | 87.5 [50 to 100] | 50 [0 to 100]
  Day 90: 2x per day prescription: number analyzed (Participants) | 10 | 3
  Day 90: 2x per day prescription | 25 [0 to 100] | 0 [0 to 0]
  Day 90: 4x per day prescription: number analyzed (Participants) | 9 | 15
  Day 90: 4x per day prescription | 50 [0 to 75] | 25 [0 to 100]
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = .002, generalized linear mixed model — The results listed here are for the main effect of time. Please see Analyses 2-3 for the main effects of time and prescription and Analyses 4-6 for interactions; Slope = -0.01 — The analyses are modeling lower adherence
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.07, generalized linear mixed model — The results listed here are for the main effect of group. Please see Analyses 1 and 3 for the main effects of time and prescription and Analyses 4-6 for interactions; Slope = -0.16 — The analyses are modeling lower adherence
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = .69, generalized linear mixed model — The results listed here are for the main effect of prescription. Please see Analyses 1-2 for the main effects of time and group and Analyses 4-6 for interactions; Slope = 0.43 — The analyses are modeling lower adherence
Statistical Analysis 4: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.37, generalized linear mixed model — The results listed here are for the time x group interaction. Please see Analyses 1-3 for the main effects of group, time and prescription and Analyses 5-7 for other interactions; Slope = 0.02 — The analyses are modeling lower adherence
Statistical Analysis 5: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.12, generalized linear mixed model — The results listed here are for the prescription x group interaction. Please see Analyses 1-3 for the main effects of group, time and prescription and Analyses 4 and 6 for other interactions; Slope = -1.14 — The analyses are modeling lower adherence
Statistical Analysis 6: Comparison: Pictorial Asthma Action Plan; The reference groups for this analysis is the 2x per day group; Test type: Superiority; p = 0.006, generalized linear mixed model — The results listed here are for the time x PAAP group x prescription interaction. Please see Analyses 1-3 for the main effects of group, time and prescription and Analyses 4-5 for interactions; Slope = 0.01 — The analyses are modeling lower adherence
Statistical Analysis 7: Comparison: Written Asthma Action Plan; The reference group for this analysis is 2x per day group; Test type: Superiority; p = 0.006, generalized linear mixed model — The results listed here are for the time x WAAP group x prescription interaction. Please see Analyses 1-3 for the main effects of group, time and prescription and Analyses 4-5 for interactions; Slope = 0.04 — These analyses are modeling lower adherence

5. Primary Outcome: Lung Function-FEV1
Description: Lung function was assessed using spirometry outcome of Forced Expiratory Volume (FEV1),
Time Frame: Measured at three time points over 6 months; baseline, 3- and 6-month follow-up.
Population: The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., equipment difficulties).
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1 value
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 23
percentage of predicted FEV1 value
  3 Month Assessment: number analyzed (Participants) | 15 | 13
  3 Month Assessment | 2.60 (1.07) | 2.39 (0.62)
  6 Month Assessment: number analyzed (Participants) | 13 | 11
  6 Month Assessment | 2.68 (0.98) | 2.66 (0.71)
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.18, multiple linear regression. — [p-value comment as in outcome 1, analysis 1]; Slope = 0.08
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.71, multiple linear regression. — [p-value comment as in outcome 1, analysis 2]; Slope = -0.09
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.96, multiple linear regression. — The results listed here are for the time x group interaction. Please see Analyses 1 and 2 for the main effects of time and group; Slope = 0.007

6. Primary Outcome: Lung Function- FEF 25-75
Description: This data is gathered from a spirometry test. FEF 25-75 is the air flow between 25% and 75% of forced vital capacity.
Time Frame: Measured at three time points over 6 months; baseline, 3- and 6-month follow-up.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 23
percent predicted
  3 month: number analyzed (Participants) | 12 | 13
  3 month | 2.88 (1.14) | 2.58 (0.68)
  6 month: number analyzed (Participants) | 11 | 10
  6 month | 2.76 (1.45) | 2.61 (0.60)

7. Secondary Outcome: Satisfaction With Asthma Action Plan-Caregiver
Description: Satisfaction questions were developed for this project and a final questionnaire developed. The Satisfaction questionnaire was completed by both parents and children at post-test (1 month, and 3 or 6 months). The scale included 11 questions, 5 reverse coded, on a 4 point Likert-type response scale. A mean item score was generated; higher scores indicate higher levels of satisfaction. Possible range of mean score was 0-4.
Time Frame: Measured at two time points over 6 months; 1- and 6-month follow-up.
Population: Pre-post analysis included combining 3 month and 6 month time points for outcome measures where the final time point was 3 instead of 6 months (N=6). The number of cases analyzed differed from the overall number analyzed due to missing data (e.g., attrition, incomplete measures).
Measure: Mean (Standard Deviation); unit: mean item score
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 22
mean item score
  1 Month Assessment | 3.64 (0.37) | 3.67 (0.30)
  Final (combined 3 month/6 month): number analyzed (Participants) | 20 | 18
  Final (combined 3 month/6 month) | 3.60 (0.35) | 3.68 (0.30)
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.74, multiple linear regression. — [p-value comment as in outcome 1, analysis 1]; Slope = -0.02
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.83, multiple linear regression. — [p-value comment as in outcome 1, analysis 2]; Slope = 0.02
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.03, multiple linear regression. — [p-value comment as in outcome 5, analysis 3]; Slope = -0.21

8. Secondary Outcome: Satisfaction With Asthma Action Plan-Patient
Description: Satisfaction questions were developed for this project and a final questionnaire developed. The Satisfaction questionnaire was completed by both parents and children at post-test (1 month, and 3 or 6 months). The scale included 11 questions, 5 reverse coded, on a 4 point Likert-type response scale. Items were averaged together for a mean score; higher scores indicate higher levels of satisfaction. Possible range of mean score was 0-4.
Time Frame: Measured at two time points over 6 months; 1- and 6-month follow-up.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mean item score
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
Number analyzed (Participants) | 22 | 22
mean item score
  1 Month Assessment | 3.65 (0.24) | 3.53 (0.40)
  Combined 3 month/6 month: number analyzed (Participants) | 20 | 19
  Combined 3 month/6 month | 3.77 (0.20) | 3.48 (0.34)
Statistical Analysis 1: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.08, multiple linear regression. — [p-value comment as in outcome 1, analysis 1]; Slope = 0.12
Statistical Analysis 2: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.25, multiple linear regression. — [p-value comment as in outcome 1, analysis 2]; Slope = -0.12
Statistical Analysis 3: Comparison: Pictorial Asthma Action Plan vs Written Asthma Action Plan; The reference for group for this analysis is the Pictorial Asthma Action Plan group; Test type: Superiority; p = 0.03, multiple linear regression. — [p-value comment as in outcome 5, analysis 3]; Slope = -0.21

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 year.
Description: The definition of adverse event and/or serious adverse event used to collect adverse event information in this study did not differ from the clinicaltrials.gov definition.
Arm/Group | Pictorial Asthma Action Plan | Written Asthma Action Plan
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT03187119/Prot_SAP_000.pdf